CLINICAL TRIAL: NCT04542824
Title: Safety and Preliminary Efficacy of Epcoritamab (GEN3013; DuoBody®-CD3×CD20) in Japanese Subjects With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma - A Phase 1/2, Open-Label, Dose-Escalation Trial With Expansion Cohorts
Brief Title: Trial of the Safety and Efficacy of Epcoritamab in Japanese Subjects With Relapsed or Refractory (R/R) B-Cell Non-Hodgkin Lymphoma (R/R B-NHL)
Acronym: EPCORE™ NHL-3
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT3013-04; JapicCTI-205408 (Registry Identifier: JAPIC); jRCT2080225312 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2020-08-25; First posted 2020-09-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma; Primary Mediastinal Large B Cell Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; R-CHOP protocol; Gemcitabine; Oxaliplatin; Maintenance; Lenalidomide

STUDY DESIGN:
Intervention Model Description: Part 1: Sequential Assignment
  Part 2: Parallel Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Arm 1: Epcoritamab (Experimental): In participants with DLBCL/FL.
  Interventions: Biological: Epcoritamab (monotherapy)
- Arm 2: Epcoritamab + Rituximab + Lenalidomide (Experimental): In participants with R/R FL
  Interventions: Biological: Epcoritamab; Drug: Rituximab and lenalidomide
- Arm 3: Epcoritamab + Rituximab + Cyclophosphamide+ Doxorubicin+ Vincristine + Prednisone (Experimental): In participants with previously untreated DLBCL
  Interventions: Biological: Epcoritamab; Drug: Rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone
- Arm 4: Epcoritamab + Gemcitabine + Oxaliplatin (Experimental): In participants with relapsed/refractory DLBCL
  Interventions: Biological: Epcoritamab; Drug: Gemcitabine and oxaliplatin
- Arm 5: Epcoritamab Maintenance (Experimental): In participants with FL in CR or in PR following 1L or 2L SOC treatment
  Interventions: Biological: Epcoritamab (maintenance)

INTERVENTIONS:
Biological: Epcoritamab (monotherapy) — Epcoritamab will be administered subcutaneously in cycles of 4 weeks (i.e. 28 days)
  Other Names: GEN3013; DuoBody®-CD3xCD20; EPKINLY™
  Arms: Arm 1: Epcoritamab
Biological: Epcoritamab — Epcoritamab will be administered in combination with the respective SOC chemotherapy followed by epcoritamab monotherapy.
  Other Names: GEN3013; DuoBody®-CD3xCD20; EPKINLY™
  Arms: Arm 2: Epcoritamab + Rituximab + Lenalidomide; Arm 3: Epcoritamab + Rituximab + Cyclophosphamide+ Doxorubicin+ Vincristine + Prednisone; Arm 4: Epcoritamab + Gemcitabine + Oxaliplatin
Drug: Rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone — 21-day cycles
  Other Names: R-CHOP
  Arms: Arm 3: Epcoritamab + Rituximab + Cyclophosphamide+ Doxorubicin+ Vincristine + Prednisone
Drug: Gemcitabine and oxaliplatin — 28-day cycles
  Other Names: GemOx
  Arms: Arm 4: Epcoritamab + Gemcitabine + Oxaliplatin
Biological: Epcoritamab (maintenance) — 28-day cycle for Cycle 1 and then 56-day cycle from Cycle 2 through 13
  Other Names: GEN3013; DuoBody®-CD3xCD20; EPKINLY™
  Arms: Arm 5: Epcoritamab Maintenance
Drug: Rituximab and lenalidomide — 28-day cycles.
  Other Names: R2
  Arms: Arm 2: Epcoritamab + Rituximab + Lenalidomide

SUMMARY:
The trial is an open-label, multi-center safety and preliminary efficacy trial of epcoritamab (EPKINLY™) in Japanese participants with relapsed, progressive or refractory B-cell lymphomas and Japanese participants with B-cell lymphomas that have achieved partial response (PR) or complete response (CR) following prior standard of care (SOC). The trial consists of two parts: Part 1, dose escalation (phase 1), and Part 2, expansion (phase 2).

The purpose of the dose-escalation part of the trial is to determine the maximum tolerated dose (MTD) and the recommended Phase-2 dose (RP2D), as well as to establish the safety profile of epcoritamab in Japanese participants with relapsed, progressive or refractory B-cell lymphoma and Japanese participants with B-cell lymphomas that have achieved PR or CR.

In the expansion part, additional participants will be treated with epcoritamab, at the RP2D and the purpose is to further explore and determine the safety and efficacy of epcoritamab.

Part 2 of the trial will be initiated once the RP2D has been determined in Part 1. In Part 2, epcoritamab is investigated as a monotherapy and in combination with other SOC agents.

DETAILED DESCRIPTION:
All participants in the trial will receive epcoritamab, as monotherapy or in combination with SOC. The following regimens will be investigated in Part 2:

Arm 1: epcoritamab monotherapy in relapsed/refractory (R/R) diffuse large B-cell lymphoma (DLBCL) and follicular lymphoma (FL)

Arm 2: epcoritamab + rituximab and lenalidomide (R2) in participants with R/R FL

Arm 3: epcoritamab + rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) in participants with previously untreated DLBCL with high risk features

Arm 4: epcoritamab + gemcitabine and oxaliplatin (GemOx) in participants with R/R DLBCL who either failed prior autologous hematopoietic stem cell transplantation (ASCT), or are ineligible for autologous HSCT.

Arm 5: epcoritamab maintenance in participants with FL who achieve a CR or a PR following first line (1L)/second line (2L) SOC treatment

ELIGIBILITY:
Main Inclusion Criteria:

• Must be at least 20 years of age, inclusive

• Japanese participants

• CD20 positivity at representative tumor biopsy

1. Part 1:

   * Diffuse large B-cell lymphoma (de novo or histologically transformed)
   * High-grade B-cell lymphoma
   * Primary mediastinal large B-cell lymphoma
   * Follicular lymphoma
   * Marginal zone lymphoma (nodal, extranodal of mucosa-associated lymphoid tissue, or splenic)
   * Small lymphocytic lymphoma
2. Part 2 :

   Arm 1:
   * Diffuse large B-cell lymphoma (de novo or histologically transformed)
   * Follicular lymphoma grade 1-3A
   * Relapsed or refractory disease and previously treated with at least 2 lines of systemic antineoplastic therapy including at least 1 anti-CD20 monoclonal antibody (mAb)-containing therapy.
   * Measurable disease by computed tomography (CT), magnetic resonance imaging (MRI) or positron emission tomography (PET)-CT scan

   Arm 2:

   • R/R FL grade 1, 2 or 3a, stage II, III, or IV, without evidence of transformation.
   * Previously treated with at least 1 prior anti-neoplastic agent, including anti-CD20 antibody
   * Must have a need for treatment initiation based on symptoms and/or disease burden (Groupe d'Etude des Lymphomes Folliculaires [GELF] criteria)
   * Eligible to receive R2 per investigator determination

   Arm 3:
   * One of following confirmed histologies (de novo or histologically transformed from FL or nodal marginal zone lymphoma) :

     o DLBCL, not otherwise specified (NOS)
     * "Double-hit" or "triple-hit" DLBCL
     * FL Grade 3B.
     * T-cell/histiocyte rich large B-cell lymphoma (LBCL)
   * International Prognostic Index (IPI) score ≥3
   * No prior therapy for DLBCL or FL grade 3B (G3B) other than nodal biopsy, corticosteroids, or palliative radiotherapy.
   * Eligible to receive R-CHOP per investigator determination

   Arm 4:
   * One of following confirmed histologies (de novo or histologically transformed from FL or nodal marginal zone lymphoma) including:

     o DLBCL, NOS.

     o "Double-hit" or "triple-hit" DLBCL
     * FL Grade 3B.
     * T-cell/histiocyte rich LBCL
   * Relapsed or refractory to at least one prior therapy including at least one prior anti-CD20 antibody.
   * Either failed prior autologous hematopoietic stem cell transplantation (ASCT), or ineligible for autologous hematopoietic stem-cell transplantation (HSCT)
   * Eligible to receive GemOx per investigator determination

   Arm 5:

   • History of histologically confirmed CD20+ FL Grade 1-3a without evidence of transformation.

   • In CR or PR per Lugano criteria following first-line or second-line treatment with SOC regimen, including anti-CD20 antibody, and last dose of SOC within 6 months prior to enrollment

   Main Exclusion Criteria:

   • Primary central nervous system (CNS) lymphoma or CNS involvement by lymphoma at screening

   • Participants not eligible for high dose therapy with autologous hematopoietic stem cell transplantation due to personal choice, social issues, or similar

   • Known clinically significant cardiac disease

   • Chronic ongoing infectious diseases requiring treatment (excluding prophylactic treatment)

   Exclusion criteria for Part 2, Arms 2 through 5:

   Arm 2:

   • FL Grade 3b

   • Histologic evidence of transformation to an aggressive lymphoma
   * Contraindication to rituximab or lenalidomide
   * Unwilling or unable to take aspirin prophylaxis or prophylactic anticoagulant as clinically indicated

   Arm 3:

   • Contraindication to any of the individual drugs of the R-CHOP regimen

   Arm 4:
   * Contraindication to any of the individual drugs of the GemOx regimen

   Arm 5:
   * FL Grade 3b
   * Histologic evidence of transformation to an aggressive lymphoma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Treatment-emergent Adverse Events (TEAEs) | From first dose until the end of the safety follow-up period (60 days after last dose), up to approximately 5 years
Part 1: Number of Participants with Dose Limiting Toxicities (DLTs) | DLTs are assessed during the first cycle (28 days) in each cohort
Part 2, Arm 1: Objective Response Rate (ORR) | Up to 1.5 years
Part 2, Arms 2-4: Number of Participants with DLTs | DLTs are assessed during the first cycle (28 days) in arms 2-4
Part 2, Arms 2-5: Number of Participants with TEAEs | From first dose until the end of the safety follow-up period (60 days after last dose), up to approximately 5 years

SECONDARY OUTCOMES:
Both parts: Area-under-the-concentration-time curve from Time 0 to Time of last dose (AUClast) | From first dose until treatment discontinuation, expected average of 1 year
Both parts: AUC from Time 0 to Infinity (AUCinf) | From first dose until treatment discontinuation, expected average of 1 year
Both parts: Maximum (Peak) Plasma Concentration (Cmax) | From first dose until treatment discontinuation, expected average of 1 year
Both parts: Time to Reach Cmax (Tmax) | From first dose until treatment discontinuation, expected average of 1 year
Both parts: Pre-dose (Trough) Concentrations (Cthrough) | From first dose until treatment discontinuation, expected average of 1 year
Both parts: Total Body Clearance of Drug from the Plasma (CL) | From first dose until treatment discontinuation, expected average of 1 year
Both parts: Volume of Distribution (Vd) | From first dose until treatment discontinuation, expected average of 1 year
Both parts: Elimination Half-life (t 1/2) | From first dose until treatment discontinuation, expected average of 1 year
Both parts: Number of Participants with Anti-Drug-Antibodies (ADAs) | From first dose until treatment discontinuation, expected average of 1 year
Part 2, Arm 1: Number of Participants with TEAEs | From first dose until the end of the safety follow-up period (60 days after last dose), up to approximately 5 years
Part 1 and Part 2, Arms 2-5: ORR | Up to 1.5 years
Both parts: CR Rate | Up to 1.5 years
Both parts: Duration of Response (DOR) | Up to 1.5 years
Both parts: Progression Free Survival (PFS) | Up to 1.5 years
Part 2: Duration of CR (DoCR) | Up to 1.5 years
Part 2: Time to Response (TTR) | Up to 1.5 years
Part 1 and Part 2 arm 1: Time to Next Anti-lymphoma Therapy (TTNT) | Up to 1.5 years
Both parts: Overall Survival (OS) | Up to 1.5 years

CONTACTS AND LOCATIONS:
Locations (15):
- Japan (15):
  - Tohoku University Hoaspital, Sendai, Miyagi
  - Aichi Cancer Center Hospital, Aichi
  - NHO Nagoya Medical Center, Aichi
  - National Cancer Center Hospital East, Chiba
  - Matsuyama Red Cross Hospital, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Kagoshima University Hospital, Kagoshima
  - Kyoto University Hospital, Kyoto
  - Kindai University Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Cancer Institute Hospital of JFCR, Tokyo
  - National Cancer Center Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Yamagata University Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Izutsu K, Akahane D, Toubai T, Saito T, Mishima Y, Fujisaki T, Nishikori M, Kumode T, Suehiro Y, Ishitsuka K, Conlon R, Takahashi A, D'Angelo Mansson B, Favaro E, Fukuhara N. Subcutaneous epcoritamab monotherapy in Japanese patients with relapsed or refractory follicular lymphoma: primary results of the EPCORE NHL-3 trial. Leuk Lymphoma. 2025 Oct;66(10):1913-1921. doi: 10.1080/10428194.2025.2525983. Epub 2025 Jul 9. PMID 40632620